CLINICAL TRIAL: NCT06111183
Title: Phase-2, Multi-centre, Prospective, Randomized, Standard-of-care Plus Placebo-controlled, Patient and Central Evaluator Blinded, Parallel Arm, Clinical Study to Evaluate Safety, Tolerability and Efficacy of the AUP1602-C as Treatment for Non-healing Neuro-ischemic DFU
Brief Title: Evaluation of AUP12602-C as New Topical Treatment for DFUs (DIAMEND STUDY)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurealis Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT-W-CLI-2022-04
Record Dates: First submitted 2023-10-09; First posted 2023-11-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This phase 2 study is patient and central evaluator (of wound images) blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AUP1602-C (Experimental): AUP1602-C is administered topically during the treatment period.
  Interventions: Biological: AUP1602-C
- Placebo (Placebo Comparator): Placebo is administered topically during the treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AUP1602-C — AUP1602-C is topically applied on chronic wounds and covered by wound dressing.
  Arms: AUP1602-C
Other: Placebo — Placebo is topically applied on chronic wounds and covered by wound dressing.
  Arms: Placebo

SUMMARY:
This is a phase 2 study performed in diabetic foot ulcer (DFU) patients with chronic non-healing, neuro-ischemic wounds to investigate the safety, tolerability and efficacy of AUP1602-C.

DETAILED DESCRIPTION:
This is a phase 2 multi-centre, parallel arm, patient and central evaluator-blinded, randomized, SoC plus placebo-controlled study of the RP2D of AUP1602-C performed in DFU patients with non-healing wounds. The RP2D of AUP1602-C derived from phase 1 study is 2.5 x 10E8 CFU/cm2 ulcer area and is used in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 and above
2. Patients with DM of type 1 or 2 having a glycosylated haemoglobin (HbA1c) of ≤ 11.0% OR 97.0 mmol/mol OR 14.9 mmol/l at randomization undergoing therapy for glycaemic control using available diabetes drugs including insulin
3. Patients with at least one DFU that fulfils all the following criteria:

   * Non-healing target ulcer defined as ≤ 20.0% reduction in area in response to SoC during the 2-weeks run-in period,
   * Duration: ≥ 4 weeks and ≤ 12 months at screening visit 1,
   * Located either in the plantar or on the dorsum of foot, or at or below the ankle,
   * Ulcer is accessible for administration of IMP and can be completely covered by the primary and secondary dressings,
   * Full-thickness, not involving bone or joints (i.e., University of Texas classification Grade 1A, 1C, 2A, 2C)(5),
   * No clinical signs of active wound infection defined by IDSA/IWGDF criteria(6) or clinical evidence osteomyelitis at randomization (V1),
   * Area of the target ulcer between 1.0-10.0 cm2 after debridement at randomization (V1)
   * Ulcer and periwound tissue suitable for application of film dressings (i.e., no contraindications and sufficient periwound space to hold the dressing).
4. Patients with more than one ulcer will be included if ulcers are separated by a minimum of 2.0 cm healthy tissue. The largest ulcer fulfilling the inclusion criteria will be selected for the investigational treatment.
5. Patients with either an ankle brachial index (ABI) ≥ 0.7 OR a toe-brachial index (TBI) ≥ 0.5, AND a toe systolic pressure of at least 50.0 mmHg (or ankle systolic pressure of at least 70.0 mmHg if toe-pressure is not measured) on the foot with the target ulcer.
6. Revascularized patients with an ulcer fulfilling the inclusion criteria can be included 3.0 months after the procedure.
7. Patients with an assessment of the baseline level of neuropathy in the lower limb where the target ulcer is located.
8. Patients must be willing to wear off-loading footwear, while ambulating, for the period requested by the Investigator.
9. A woman of childbearing potential (WOCBP) must have a negative serum pregnancy test at the time of screening after sign the informed consent and a negative pregnancy dip-stick test at baseline (before starting treatment).
10. Females of childbearing potential must agree to use a highly effective contraceptive measure (methods that can achieve a failure rate of less than 1% per year when used consistently and correctly) , throughout the study. / Male patients who are biologically capable of having children must agree to apply at least two methods of contraception including male barrier protection throughout the study.
11. Patients who understand and are willing to comply with study procedures and give written informed consent prior to enrolment in the study or initiation of study procedures.

Exclusion Criteria:

1. Participating in another clinical study or treatment with another investigational product and/or medical device in the 30 days prior to inclusion in the study or within the 5 half-lives of the investigational product, whichever is longer.
2. Current or previous (within 30 days prior to start of run-in period) treatment of target ulcer with a treatment that could interfere with wound healing/IMP such as biological agents, growth factors, skin equivalents/substitutes (e.g., Regranex®, Apligraf®, or Dermagraft®), keratinocytes, platelet-rich-plasma, collagen products, blood products, placental products, oxygen therapy, topical steroids.
3. Current or previous (within 1 week prior to first IMP (AUP1602-C or placebo) dosing) treatment with active wound care agents (e.g., local/topical antibiotics OR antibacterials such as silver, iodine, chlorhexidine) OR systemic antibiotics for any indication.
4. Current or previous (within 2 weeks prior to first IMP (AUP1602-C or placebo) dosing) use of corticosteroids and immunosuppressants. Treatment with immunosuppressive agents with known therapeutic effects longer than 2 weeks may be considered as exclusion and should be consulted with Medical Monitor/Sponsor.
5. Known hypersensitivity to any of the components of AUP1602-C or placebo
6. Ulcer of University of Texas Grade ≥ 3, with deep abscess, sinus track, necrosis or gangrene that cannot be removed by debridement.
7. Target ulcers with excessive exudation requiring more than one dressing change within 24-hrs.
8. Target ulcers with clinically significant periwound skin maceration.
9. Target ulcer with known or suspected active infection, which requires antimicrobials. Any antibiotic therapy must be completed or discontinued within 1 week prior to first IMP (AUP1602-C or placebo) dosing.
10. Target ulcers requiring urgent vascular surgical interventions.
11. Target ulcer other than non-healing DFU fulfilling inclusion criteria (e.g., including, but not limited to, pressure ulcers, burn wounds).
12. Serum creatinine level of > 3.0 times the upper limit of normal (ULN).
13. Prior radiation therapy (within 6 weeks prior to first IMP (AUP1602-C or placebo) dosing) of any part of the foot/leg bearing the target ulcer under study or total body irradiation.
14. Sickle-cell diseases, Reynaud's, or other peripheral vascular disease including venous leg ulcers or any vasculitic ulcer irrespective of the cause will be excluded.
15. Active or unstable Charcot deformity of the study foot (i.e., foot is erythematous, warm, oedematous, and is actively remodelling).
16. Patients with other reasons for wound healing disturbances: e.g., bleeding disorders, vitamin K deficiency, hypocalcaemia, major immune deficiencies.
17. Active malignant disease of any kind except for basal cell carcinoma (of the skin) not co-located with the target ulcer. A patient, who has had a malignant disease in the past, completed treatment and is currently disease-free and not on active treatment for at least 3 months, may be considered for study entry. Cancer therapies with known therapeutic effects longer than 3 months may be considered as exclusion and should be consulted with Medical Monitor/Sponsor.
18. Haemoglobin of less than 8.5 g/dL
19. Liver transaminase & total bilirubin levels greater than 3 times ULN.
20. Patients receiving haemodialysis or continuous ambulatory peritoneal dialysis (CAPD) therapy.
21. Positive for hepatitis B or C virus (HBV, HCV), or human immunodeficiency virus (HIV) (serology test results up to 3 months prior signing ICF accepted).
22. Patients with confirmed active infection with SARS-CoV-2 and related disease (COVID-19) at Baseline (V1) prior to first administration of trial medication.
23. Planned major surgery during the run-in, treatment and post-treatment efficacy and safety follow-up period of the study.
24. Known abuse of alcohol, drugs, or medical products. Tobacco use will be allowed.
25. Previous treatment with AUP1602-C.
26. Any diagnosed unstable psychological or physical condition including major organ failure that could interfere with compliance.
27. Myocardial infarction diagnosed within 1 month prior to start of run-in period.
28. White Blood Cells (WBC) < 3.0 X 109 cells/L；> 12.0 X 109 cells/L
29. Albumin < 2.5 g/dL (or total protein < 4.0 g/dl).
30. The patient has any other factor/reason which may, in the opinion of the Investigator, compromise participation and/or follow-up in the study.
31. Pregnant or lactating woman at the time of signing the informed consent and prior to first IMP (AUP1602-C or placebo) dosing.
32. Close affiliation with the Investigator (e.g., a close relative, financially dependent on the investigational site) or patient who is an employee of the Sponsor's company.
33. Patients who are institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systematic adverse events (AEs) | 6 weeks
  Incidence of local and systematic adverse events (AEs) for repeatedly administered AUP1602-C and of the placebo control arm.
Incidence of Wound Closure | 20 weeks
  Proportion of patients with a target ulcer achieving complete wound closure

SECONDARY OUTCOMES:
To evaluate the effect size of the efficacy parameters for AUP1602-C and placebo control arm in DFU patients | 20 weeks
  * Percentage of wound area reduction
  * Percentage of wound volume and depth reduction
To evaluate the effect size of the efficacy parameters for AUP1602-C and placebo control arm in DFU patients | 20 weeks
  * Time to complete wound closure
  * Time to >50% wound area reduction
  * Time to >75% wound area reduction
To evaluate the effect size of the efficacy parameters for AUP1602-C and placebo control arm in DFU patients | 20 weeks
  * Proportion of patients with complete wound closure
  * Proportion of patients with a >50% wound area reduction
  * Proportion of patients with a >75% wound area reduction
  * Proportion of patients with a target ulcer recurrence
To evaluate the effect of the RP2D and selected treatment schedules on the percentage of wound area reduction in DFU patients | 20 weeks
  • Percentage of wound area reduction
To evaluate the effect of the RP2D and selected treatment schedules on the percentage of wound area reduction in DFU patients | 20 weeks
  * Time to complete wound closure
  * Time to >50% wound area reduction
  * Time to >75% wound area reduction
To evaluate the effect of the RP2D and selected treatment schedules on the percentage of wound area reduction in DFU patients | 20 weeks
  * Proportion of patients with complete wound closure
  * Proportion of patients with a >50% wound area reduction
  * Proportion of patients with a >75% wound area reduction
To evaluate the effect of the RP2D and selected treatment schedules long-term healing in DFU patients | 20 weeks
  • Proportion of patients with complete wound closure
To evaluate the effect of the RP2D and selected treatment schedules ulcer recurrence in DFU patients | 20 weeks
  • Proportion of patients with a target ulcer recurrence
Changes in Quality of Life according to EQ-5D-5L | 20 weeks
  Change from baseline in health-related quality is assessed according to EuroQoL-5 Dimensions (EQ-5D-5L) patient quesionnaire. Five single-item dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) are assessed. Result of the questionnaire is scored from 0 (worst health imaginable) to 100 (best health imaginable).
Changes in Quality of Life according to DLQI | 20 weeks
  Change from baseline in health-related quality is assessed according to Dermatology Life Quality Index (DLQI). It consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score will be calculated as the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life.
Changes in pain assessment according to VAS | 20 weeks
  Change from baseline in patient's pain intensity according to a numerical Visual Analog Scale (VAS) ranging from 0 = no pain to 10= worst imaginable pain.
Incidence of target ulcer related hospital visits | 20 weeks
  * Number of target ulcer related hospital visits
  * Number of patient-days of hospitalization due to complications related to target ulcer
  * Number of patient-days of target ulcer related antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (2):
  - Institut für Diabetesforschung Muenster GmbH, Münster
  - Hauärztliche und Diabetologische Praxis, Pirna
- Italy (4):
  - Ospedale San Donato, Arezzo
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AOU Pisana - Ospedale S. Chiara, Pisa
  - Ospedale S. Jacopo Pistoia, Diabetologia e Diabetic foot unit Aziendale, Pistoia
- Poland (4):
  - Mikomed, Lodz
  - Med-Polonia SP. Z O.O., Poznan
  - PODOS Klinika Leczenia Ran Podema sp. z o.o., Warsaw
  - Lecran Centrum Opieki Nad Ranami, Wroclaw

IPD SHARING:
Plan to Share IPD: No